CLINICAL TRIAL: NCT04146415
Title: Diagnosis of Cardiac Amyloidosis With 99mTc-PYP; Comparison Between Planar Imaging, SPECT/CT and Cardiac-dedicated CZT Camera
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TASMC-18-ES-0042-CTIL
Record Dates: First submitted 2019-10-29; First posted 2019-10-31 (Actual); Last update posted 2019-11-06 (Actual); Status verified 2019-11

CONDITIONS: Cardiac Amyloidosis
MeSH Terms: conditions — Amyloid Neuropathies, Familial | interventions — Tomography, Emission-Computed, Single-Photon

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cardiac amyloidosis patients (Experimental)
  Interventions: Diagnostic Test: Spect scan with mTc99-PYP

INTERVENTIONS:
Diagnostic Test: Spect scan with mTc99-PYP — . About forty-five minutes after the injection mTc99-PYP , flanner and SPECT-CT mappings will be performed and then the patient will move to the CZT camera and undergo another photograph.

SUMMARY:
1. Patients will undergo clinical and laboratory assessment, as well as imaging tests, at the discretion of the attending cardiologist and will be referred at their discretion to perform cardiac mapping using 99mTc-PYP.
2. On the day of the examination, the examiner will be admitted to the Office of Nuclear Medicine and will be admitted to administrative. Before conducting the test, the subject will undergo a brief interview by a physician, receive an explanation of the study and, if agreed, sign an agreement to perform a further examination on the CZT camera.
3. The patient will, as is customary, be installed on Vanflon 22 G periphery, through which a 15 millikiric (mCi) of

ELIGIBILITY:
Inclusion Criteria:

A. Patients undergoing "cardiac amyloidosis clinic" at Tel Aviv Medical Center and there is a clinical suspicion of having cardiac amyloidosis.

B. Patients who performed will be referred for mapping using 99mTc-PYP and sign a consent form to take another photograph, under the cardiac-dedicated CZT camera

Exclusion Criteria:

1.None

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-11-01 (Estimated); Primary Completion 2019-11-30 (Estimated); Study Completion 2020-08-01 (Estimated)

PRIMARY OUTCOMES:
Patients who preformed mTc99-PYP for cardiac amyloidosis imaging. | 1 year
  Evaluation of cardiac amyloidosis imaging with mTc99-PYP cardiac-dedicated CZT camera

IPD SHARING:
Plan to Share IPD: Undecided